CLINICAL TRIAL: NCT02740738
Title: Preoperative Pain Threshold and Rapid Recover Programs in Total Joint Arthroplasty
Brief Title: Preoperative Pain Threshold and Rapid Recover Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00069521
Record Dates: First submitted 2016-03-16; First posted 2016-04-15 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Knee Arthritis; Hip Arthritis
Keywords: Knee Arthroplasty; Hip Arthroplasty
MeSH Terms: interventions — Muscle Strength Dynamometer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wagner Pain Algometer — applied at a 90 degree angle to the skin at a constant rate of 10kPa/s to minimize the impact of the examiner's reaction time on recorded pain thresholds
Device: Dynamometer — Dominant Hand Grip strength measured by the average of 3 attempts

SUMMARY:
To investigate the association between grip strength and preoperative pain threshold as measured by pressure algometer and validated pain outcome surveys.

DETAILED DESCRIPTION:
A minimum of 200 patients, 100 hip and 100 knee arthroplasty participants, will be recruited for this study. Preoperatively, patient pain threshold will be recorded both objectively (Pressure algometer) and subjectively (brief pain inventory). In terms of location, objectively this will be tested during the preoperative visit in clinic by the approved, trained research staff, as well as the subjective brief pain inventory.

Objective pain measure: Pressure algometer will be obtained in the standard fashion as follows: the probe is applied at a 90 degree angle to the skin at a constant rate of 10kPa/s to minimize the impact of the examiner's reaction time on recorded pain thresholds. The participant is instructed by the measurer to say "stop" when the sensation of pressure became the very first sensation of pain. There will be three spots to test patients, one for familiarity of the testing and the other 2 for data collection.

1. This is initially performed once on ipsilateral the tibialis anterior as a "warm up."
2. Then 3 measurements are taken on the operative medial epicondyle (for TKA) or ipsilateral lateral iliac crest (for THA) and averaged for the official score.
3. Lastly, three measurements are also taken on the contralateral olecranon to measure systemic pain sensitivity. If the contralateral elbow has had prior surgery or active bursitis, the ipsilateral elbow will be used. Of important note, the algometer has a max force lock out of 100N to prevent any harm to the patient.
4. Dominant Hand Grip strength measured by the average of 3 attempts on a Dynamometer.

Subjectively, the brief pain inventory is a validated pain outcome measure which will be filled out by the participant during their preoperative clinic visit.

Postoperative, the study team will ask the participant at the 6 week mark:

1. How many and what kind of opiates did the participant require?
2. How many days did the participant require opiates?
3. Did the participant require a refill? a. If so, did the participant have this filled in clinic preemptively or place a phone call to the office?

ELIGIBILITY:
Inclusion Criteria:

* any participant undergoing elective primary total knee arthroplasty or total hip arthroplasty
* Participants of the following investigators will be approached: Bolognesi, Wellman, Attarian, and Seyler

Exclusion Criteria:

* previous hip or knee surgery in the operative joint

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-03; Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Inpatient length of stay in days | 1-3 on days average
  amount of time in hospital
pain control average visual analogue scale 1 - 10 of hospital stay | 1-3 days on average
  averaging the subjective pain control
physical therapy performance on the first day after surgery | post op day 1
  distance walked in feet on post op day 1
discharge location placement | 1 - 3 days on average
  home, rehab or nursing facility

SECONDARY OUTCOMES:
Outpatient narcotic pill consumption | 6-week from surgery
  narcotic equivalents consumed by patient in morphine equivalents. we will convert all medicine to the standard unit
Outpatient narcotic consumption refill needed | 6-week from surgery
  need for refill prescription, yes or no
Outpatient narcotic consumption multiple refills needed | 6-week from surgery
  number of refills needed requiring provider time outside of scheduled appointment

OTHER OUTCOMES:
Complications short term after surgery | 6-week from surgery
  Inpatient complications while in the hospital
Complications long term after surgery | surgery to 1yr postoperative
  Outpatient complications seen after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wellman, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Plaza Page Road, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No